CLINICAL TRIAL: NCT03637985
Title: Exercise and Menopausal Hypertension
Brief Title: Effect of 12 Weeks of Resistive Exercises Versus Aerobic Exercises in Overweight Hypertensive Postmenopausal Women
Acronym: exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Ebrahim El Refaye, Assistant Professor of physical therapy for women's health, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CairoU89
Record Dates: First submitted 2018-08-07; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Exercise
Keywords: resistive exercises; aerobic; Menopause; hypertension
MeSH Terms: conditions — Motor Activity; Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The allocation was concealed in sequentially numbered opaque envelopes by a blinded and an independent research assistant and selected 69 individuals randomly into the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- resistive exercise (Experimental): resistive exercises using elastic band(Thera Band) Sets were at moderate intensity, 8-10 repetitions for every motion for 12 weeks
  Interventions: Device: resistive exercise
- Aerobic exercise (Experimental): Aerobic exercise in form of treadmill walking for 45 minutes for 12 weeks
  Interventions: Device: aerobic exercise in form of treadmill walking

INTERVENTIONS:
Device: resistive exercise — resistive exercise by elastic band for 12 weeks
  Arms: resistive exercise
Device: aerobic exercise in form of treadmill walking — aerobic exercise in form of treadmill walking for 12 weeks
  Arms: Aerobic exercise

SUMMARY:
Sixty postmenopausal women participated in this study from gynecological outpatient clinic, at Al-Zahra universal Hospital, Al Azhar University, and Cairo. They were first diagnosed to be hypertensive in their early postmenopausal period .Their blood pressure ranged between 140/90mmHg to 170/105mmHg, their ages ranged from 50 to 60 years and their body mass index ranged from 30:35 kg/m2.

DETAILED DESCRIPTION:
The participants were divided randomly according to closed envelop into three equal groups in number: Group A (RE) consisted of twenty women who participated in the resistive exercise program. Group B (AE) group: consisted of twenty women who participated in an aerobic exercise program. All patients in both groups (A & B) participated in the exercises three times per week for twelve weeks and every session lasted for 45 min and continues their antihypertensive medication

ELIGIBILITY:
Inclusion Criteria:

* All women diagnosed as essential hypertension.
* All women must be in their early postmenopausal period

Exclusion Criteria:

* Lesion to higher centers leading to hypertension (embolism)
* any cardiovascular disease
* premature menopause
* surgical menopause
* severe hypertension
* diabetic
* under treatment of hormonal therapy.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Assessment of changes in the systolic blood pressure | 12 weeks
  using the mercury column sphygmomanometer

SECONDARY OUTCOMES:
Assessment of changes in the diastolic blood pressure | 12 weeks
  using the mercury column sphygmomanometer

CONTACTS AND LOCATIONS:
Overall Officials: ghada E elrefaye, Professor, Principal Investigator — Assistant professor of physical therapy for women's health
Locations (1):
- Al Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
a randomized controlled trial to determine and compare effect of 12 weeks of resistive exercises versus aerobic exercises in treatment of postmenopausal hypertension
Supporting Information: SAP, ICF, CSR
Time Frame: from 1 September 2017 to 1 August 2018